CLINICAL TRIAL: NCT04033913
Title: What Are the Criteria for the Patient's Choice of Sel-catheterization Catheter
Status: Completed | Type: Observational
Sponsor: Gérard Amarenco (Other)
Responsible Party: Sponsor-Investigator, Gérard Amarenco, Head of Neuro-Urology department, Tenon Hospital, Pierre and Marie Curie University
Organization: Pierre and Marie Curie University (Other)
Other Study IDs: GRC-01 GREEN
Record Dates: First submitted 2019-07-20; First posted 2019-07-26 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Intermittent Urethral Catheterization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patient learning self-catheterization: Patients who have successfully perform self-catheterization during a day hospital in a neuro-urology department complete a questionnaire validated by experts on the different criteria that guided the final choice of the catheter
  Interventions: Other: Self questionnaire

INTERVENTIONS:
Other: Self questionnaire — Patients who have successfully perform self-catheterization complete a self questionnaire on the importance of each criterion in choosing the catheter they have made.

SUMMARY:
The aim of this study is to evaluate which are the most important criteria guiding the choice of the catheter for the patient to perform clean intermittent self catheterization.

DETAILED DESCRIPTION:
Management of voiding dysfunction has been revolutionized by the practice of clean intermittent self-catheterization (CISC) described by Lapides. It is nowadays the gold standard for the treatment of urinary retention in neurogenic bladders. But increasingly, CISC is prescribed to patients with non-neurogenic lower urinary tract symptoms (LUTS). Several studies have demonstrated an improvement in quality of life in patients under CISC. There are several indications for CISC in older adults, either in neurological condition (myelopathy following neck osteoarthritis, lumbar spinal stenosis, multiple sclerosis (MS), etc…) or not (bladder outlet obstruction, underactive detrusor, etc…).

The arrival of hydrophilic catheters has revolutionized management, reducing the risk of traumatic and infectious complications and facilitating their use. Many catheters are now available, and the choice of catheter may depend on different factors: grip disorder, ease of use, design and packaging, discomfort or pain when testing a specific material, specific anatomical conditions (male Tiemann or olive tip), longer catheter length in case of imperfect emptying, explanations given on how to use the catheter... Thus, if the doctor and the nurse involved in the patient's therapeutic education in self-catheterization will guide the choice of the catheter according to medical criteria and the patient's physical capacities, the patient remains an active participant in the choice of the model. Making the patient an actor and decision-maker can also improve adherence to treatment.

The aim of this study is to evaluate which are the most important criteria guiding the choice of the catheter for the patient.

In this study, the investigators develop a questionnaire based on expert meetings and literature review of the criteria that guide the choice of the catheter.

Five areas are explored: catheter design, catheter length, comfort of using the catheter, nurse's explanations, easy to transport and dispose of the catheter.

The importance of each criterion is rated by a 4-level likert scale (strongly disagree, somewhat disagree, somewhat agree, strongly agree) and patient have to report the most important criterion for the choice of the catheter.

Number of types of catheter showed and tried are reported, and if they chose the first, second, are two types of catheter. The questionnaire is completed at the end of a day hospital to learn to perform CISC

Data collected are:

* Age
* Sex
* Etiology of urinary disorders
* Score of the Pencil and Paper Test
* Functional Independence Measure score
* Nine Hold Peg Test over 18
* "Tinetti Mobility Test" score
* sensory hand problems assessed by Weber test

Statistical analyses will be performed with the R software for Windows (Rx64 3.2.3, R Foundation for Statistical Computing, Vienna, Austria). Descriptive data will be presented as means with standard deviation for continuous data and as medians with range for ordinal data and data not normally distributed.

Differences between the choosing criterion and the patients' characteristics will be assessed using analysis of variance or Chi2 tests. A p value of less than 0.05 will be considered statistically significant.

This study was approved by the local ethics review board.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients who have successfully perform self-catheterization during a day hospital in a neuro-urology department

Exclusion Criteria:

* patient who does not speak French
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients who have successfully perform self-catheterization during a day hospital in a neuro-urology department
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-08-10 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
The criterion of the created questionnaire for the choice of the catheter designated by the patient as the most important (rate of patients who identified each criterion as the most important) | 1 day
  patients must identify the most important criterion among the 5 proposed in the questionnaire created: catheter design; catheter length; comfort to handle the catheter; nurse's explanations; discretion for transport and disposal of the catheter.
  Only one answer is accepted.

SECONDARY OUTCOMES:
Importance for the choice of catheter of each of the 5 criteria of the questionnaire created, using a 4-level likert scale | 1 day
  the importance of each criterion (catheter design; catheter length; comfort to handle the catheter; nurse's explanations; discretion for transport and disposal of the catheter) is rated by a 4-level likert scale (strongly disagree, somewhat disagree, somewhat agree, strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Amarenco, PhD, Principal Investigator — Sorbonne Université, GRC 001, GREEN, AP-HP, Hôpital Tenon, Paris, France
Locations (1):
- department of Neuro-Urology, Hôpital Teno, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided